CLINICAL TRIAL: NCT03823170
Title: Effectiveness of Laser Therapy Associated With Fluoride Therapy in Hypomineralized Teeth Desensibilization: Randomized Clinical Trial
Brief Title: Laser Therapy and Flouride Therapy in Desensibilization Hypomineralized Teeth
Acronym: LTAFTIDHT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Ceuma (Other)
Collaborators: Fundação de Amparo à Pesquisa e Desenvolvimento Científico do Maranhão (Unknown)
Responsible Party: Principal Investigator, Meire Coelho Ferreira, Study Director, Universidade Ceuma
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MCCF-230784-RM
Record Dates: First submitted 2019-01-28; First posted 2019-01-30 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Hypomineralization Molar Incisor
Keywords: hypomineralization molar incisor; Child; Laser Therapy; Tooth Sensitivity
MeSH Terms: conditions — Molar Hypomineralization; Dentin Sensitivity | interventions — Laser Therapy

STUDY DESIGN:
Intervention Model Description: Groups: treatment with laser therapy (Group 1); treatment with fluorotherapy (Group 2) and treatment with laser therapy and fluorotherapy (Group 3).
Who Masked: Outcomes Assessor
Masking Description: The researcher who will evaluate the treatments through the syringe test will be masked as to the type of treatment performed in each patient. The investigator responsible for the treatment and the patient will not be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Laser therapy (Experimental): The low-power, infrared (808nm wavelength) diode laser with a power of 100mW (Therapy EC, DMC) will be used. The mode of irradiation is punctual, in contact and perpendicular to the dental surface. Three points on the crown of multiradicular teeth (mesial and distal of the cervical region and central part of the tooth lesion) and two points on the crown of unirradicular teeth (central point of the cervical region and central part of the tooth lesion) will be irradiated for 10s per point , 1J per point, with a 72-hour interval between treatment sessions. The distance between the irradiation points will be about 2 mm. The tip of the laser equipment will be positioned perpendicular to the application site.
  Interventions: Radiation: Laser therapy
- Fluorotherapy (Active Comparator): The treatment will be carried out with the application of fluoride varnish (Duraphat), with the aid of a microbrush. After the application, water will be dripped onto the applied varnish in order to promote its drying. Fluorotherapy will be performed once a week, totaling 4 sessions.
  Interventions: Procedure: Fluorotherapy
- Laser therapy and fluorotherapy (Experimental): The teeth will be treated first with the laser (same specifications as Laser therapy), followed by application of fluoride varnish (same specifications as Fluorotherapy).
  Interventions: Combination Product: Laser therapy and Fluorotherapy

INTERVENTIONS:
Radiation: Laser therapy — The low-power, infrared (808nm wavelength) diode laser with a power of 100mW will be used. The mode of irradiation is punctual, in contact and perpendicular to the dental surface. Three points on the crown of multiradicular teeth (mesial and distal of the cervical region and central part of the tooth lesion) and two points on the crown of unirradicular teeth (central point of the cervical region and central part of the tooth lesion) will be irradiated for 10s per point , 1J per point, with a 72-hour interval between treatment sessions. The distance between the irradiation points will be about 2 mm. The tip of the laser equipment will be positioned perpendicular to the application site.
  Arms: Laser therapy
Procedure: Fluorotherapy — The treatment will be carried out with the application of fluoride varnish, with the aid of a microbrush. After the application, water will be dripped onto the applied varnish in order to promote its drying. Fluorotherapy will be performed once a week, totaling 4 sessions.
  Arms: Fluorotherapy
Combination Product: Laser therapy and Fluorotherapy — This group will be treated first with the laser (same specifications as Laser therapy), followed by application of fluoride varnish (same specifications as Fluorotherapy).
  Arms: Laser therapy and fluorotherapy

SUMMARY:
To investigate the efficacy of laser therapy associated with fluorotherapy in the desensibitization of hypomineralized teeth in children 8 to 12 years of age. A randomized blinded clinical trial will be conducted. The instruments used will be a questionnaire general, clinical examination, dental air syringe (evaluation of dental sensitivity) and visual analogue scale (evaluation of the magnitude of dental sensitivity). Teeth with hypomineralization molar-incisor (HMI) and the results of sensitivity and magnitude of dental pain before and after the treatments will be recorded in a clinical record. The study groups will be: treatment with laser therapy (Group 1); treatment with fluorotherapy (Group 2) and treatment with laser therapy and fluorotherapy (Group 3).

DETAILED DESCRIPTION:
A blinded randomized clinical trial will be conducted. The study will be conducted with children attending the Pediatric Dentistry Clinic of the Florence Institute's undergraduate course, in São Luís, Maranhão, Brazil. As inclusion criteria, children from 8 to 12 years of age will be adopted, with at least one first permanent or incisive erupted incisor (with occlusal / incisal surface free of gingiva) present in the oral cavity and presenting sensitive hypomineralization lesions. Exclusion criteria will be children with enamel malformations linked to syndromes, with dental fluorosis, enamel hypoplasia or with imperfect amelogenesis, teeth with loss of structure dental and carious lesions, children in orthodontic treatment, children with cognition problems, children who used any type of analgesic / anti-inflammatory medication before treatment, children undergoing desensitizing treatment in the last 3 months, children with behavioral problems and children with occlusal problems such as tightening and bruxism.

The instruments of data collection will be a general questionnaire (demographic, socioeconomic and etiological factors for HMI), clinical examination for diagnosis of HMI, dental sensitivity test with air syringe and visual analogue scale (to assess the magnitude of pain). In a clinical file will be recorded the teeth with HMI, the result of the sensitivity test and magnitude of dental pain before and after treatments. The general questionnaire will be answered by the parents / guardians. In cases of incomplete questionnaires, parents / guardians will be contacted by telephone.

The diagnosis of HMI will be performed according to the criteria proposed by the European Academy of Child Dentistry (WEERHEIJM et al., 2003). The researcher will be calibrated for the application of the questionnaire and for the diagnosis of HMI lesions.

The study groups will be: treatment with laser therapy (Group 1); treatment with fluorotherapy (Group 2) and treatment with laser therapy and fluorotherapy (Group 3). For the treatment of group 1, the low-power, infrared (808nm wavelength) diode laser with a power of 100mW will be used. The mode of irradiation is punctual, in contact and perpendicular to the dental surface. Three points on the crown of multiradicular teeth (mesial and distal of the cervical region and central part of the tooth lesion) and two points on the crown of unirradicular teeth (central point of the cervical region and central part of the tooth lesion) will be irradiated for 10s per point , 1J per point, with a 72-hour interval between treatment sessions. The distance between the irradiation points will be about 2 mm. The tip of the laser equipment will be positioned perpendicular to the application site. The treatment of Group 2 will be carried out with the application of fluoride varnish, with the aid of a microbrush. After the application, water will be dripped onto the applied varnish in order to promote its drying. Fluorotherapy will be performed once a week, totaling 4 sessions. Group 3 will be treated first with the laser (same specifications as Group 1), followed by application of fluoride varnish (same specifications as Group 2).

ELIGIBILITY:
Inclusion Criteria:

* Children from 8 to 12 years of age;
* At least one first permanent or incisive erupted incisor (with occlusal / incisal surface free of gingiva) present in the oral cavity;
* Teeth presenting hypomineralization lesions sensitive.

Exclusion Criteria:

* Children with enamel malformations linked to syndromes, with dental fluorosis, enamel hypoplasia or with imperfect amelogenesis;
* Teeth with loss of dental structure and carious lesion;
* Children in orthodontic treatment;
* Children with cognition problems;
* Children who used any type of analgesic / anti-inflammatory medication before treatment;
* Children undergoing desensitizing treatment in the last 3 months
* Children with behavioral problems;
* Children with occlusal problems such as tightening and bruxism.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2018-12-23 (Actual); Study Completion 2018-12-23 (Actual)

PRIMARY OUTCOMES:
Dental sensitivity | 1 month after the onset of treatment
  The dental sensitivity will be evaluated with air from the dental syringe.

CONTACTS AND LOCATIONS:
Overall Officials: Meire C. Ferreira, PhD, Study Director — Uniceuma; Rosyara SC Muniz, DDS, Principal Investigator — Uniceuma
Locations (1):
- Josue Montello, Universidade Ceuma, São Luís, Maranhão, Brazil

REFERENCES:
- [Result] Ghanim A, Silva MJ, Elfrink MEC, Lygidakis NA, Marino RJ, Weerheijm KL, Manton DJ. Molar incisor hypomineralisation (MIH) training manual for clinical field surveys and practice. Eur Arch Paediatr Dent. 2017 Aug;18(4):225-242. doi: 10.1007/s40368-017-0293-9. Epub 2017 Jul 18. PMID 28721667
- [Result] Lopes AO, Eduardo Cde P, Aranha AC. Clinical evaluation of low-power laser and a desensitizing agent on dentin hypersensitivity. Lasers Med Sci. 2015 Feb;30(2):823-9. doi: 10.1007/s10103-013-1441-z. Epub 2013 Oct 4. PMID 24197517
- [Result] Aranha AC, Pimenta LA, Marchi GM. Clinical evaluation of desensitizing treatments for cervical dentin hypersensitivity. Braz Oral Res. 2009 Jul-Sep;23(3):333-9. doi: 10.1590/s1806-83242009000300018. PMID 19893971
- [Result] Lygidakis NA, Wong F, Jalevik B, Vierrou AM, Alaluusua S, Espelid I. Best Clinical Practice Guidance for clinicians dealing with children presenting with Molar-Incisor-Hypomineralisation (MIH): An EAPD Policy Document. Eur Arch Paediatr Dent. 2010 Apr;11(2):75-81. doi: 10.1007/BF03262716. PMID 20403301
- [Result] Ozgul BM, Saat S, Sonmez H, Oz FT. Clinical evaluation of desensitizing treatment for incisor teeth affected by molar-incisor hypomineralization. J Clin Pediatr Dent. 2013 Winter;38(2):101-5. PMID 24683770
- [Result] Palazon MT, Scaramucci T, Aranha AC, Prates RA, Lachowski KM, Hanashiro FS, Youssef MN. Immediate and short-term effects of in-office desensitizing treatments for dentinal tubule occlusion. Photomed Laser Surg. 2013 Jun;31(6):274-82. doi: 10.1089/pho.2012.3405. Epub 2013 May 15. PMID 23675985